CLINICAL TRIAL: NCT05393752
Title: Evaluation of Malnutrition Risk Assessment Tools in General Surgery.
Brief Title: Malnutrition Assessment Tools in Surgery
Acronym: MATS
Status: Completed | Type: Observational
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Konstantinos Lasithiotakis, Assisstant Professor of Surgery, University Hospital of Crete
Other Study IDs: 18981/4-11-2021
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Malnutrition; Surgery--Complications
Keywords: nutrition; malnutrition; malnutrition risk tools; nutritional assessment; surgery
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the main malnutrition risk assessment tools in patients undergoing operations of general surgery.

DETAILED DESCRIPTION:
This is a multi centre prospective observational study including patients undergoing major/major+ operation of general surgery. Patients will be interviewed by surgical trainees and their malnutrition risk will be assessed with the use of SGA, MUST, NRS, MNA-SF etc. Clinical variables and demographics will also be recorded in order to enable meaningful comparisons of malnutrition risk assessment tools in terms of serious postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients undergoing elective or emergency surgery. Urgency of emergent operations is classified as follows, according to the clinical judgment of the surgeon, regarding the maximum time a patient could wait for surgery:

  * 3.Expedited (>18 hours)
  * 2B. Urgent (6-18 hours)
  * 2A. Urgent (2-6 hours)
  * 1. Immediate (<2 hours)
* Operations involving the gastrointestinal tract
* Magnitude of operation graded by POSSUM [17,18]:

  * Major+ (examples include colonic resection abdominoperineal resection of the rectum, radical total gastrectomy, intestinal bypass, whipple resection)
  * Major (examples include adhesiolysis, stoma formation, small bowel resection, anterior resection, cholecystectomy and exploration of the bile duct)

Exclusion Criteria:

* Age <18 years
* Magnitude of operation graded by POSSUM:

  * Minor
  * Intermediate
* Inability to perform nutritional assessment
* Inability to provide informed consent

Ages: 18 Years to 108 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study including patients admitted in a surgical department during a 1-year study period, from January 2022 until January 2023 (TBReviewed)
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
serious postoperative complications | 30 days after the operation
  Complications >II according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Lasithiotakis, MD, PhD, Principal Investigator — University Hospital of Heraklion, Crete, Greece
Locations (2):
- Department of Surgery, General Hospital of Nicosia, School of Medicine, University of Cyprus, Nicosia, Cyprus
- Department of Surgery, University Hospital of Heraklion, Heraklion, Greece

IPD SHARING:
Plan to Share IPD: No